CLINICAL TRIAL: NCT07318103
Title: A Multicentre, Randomised, Double-blind, Placebo-controlled Phase II Clinical Study Evaluating the Efficacy and Safety of Injectable HRS-9057 in Patients With Heart Failure-induced Fluid Retention
Brief Title: Phase II Clinical Study of HRS-9057 Injection in Patients With Heart Failure-induced Fluid Retention
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-9057-201
Record Dates: First submitted 2025-11-21; First posted 2026-01-05 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-11

CONDITIONS: Fluid Retention Caused by Heart Failure
MeSH Terms: interventions — Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRS-9057 for injection (Experimental)
  Interventions: Drug: HRS-9057 injection set
- 5% Glucose Injection (Placebo Comparator)
  Interventions: Drug: 5% Glucose Injection

INTERVENTIONS:
Drug: HRS-9057 injection set — HRS-9057 injection set
  Arms: HRS-9057 for injection
Drug: 5% Glucose Injection — 5% Glucose Injection
  Arms: 5% Glucose Injection

SUMMARY:
Phase II clinical study of HRS-9057 injection in patients with heart failure-induced fluid retention

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years on the day of signing the informed consent, regardless of gender;
2. Hospitalised for acute heart failure within 24 hours prior to randomisation;
3. Presence of heart failure symptoms before randomisation (exertional dyspnoea, nocturnal paroxysmal dyspnoea, orthopnoea, etc.) and at least one sign of fluid retention, including: pulmonary rales on auscultation, pitting oedema of the lower limbs, pulmonary congestion confirmed by chest imaging;
4. NT-proBNP >450 pg/mL within 12 hours prior to randomisation, >600 pg/mL for patients with atrial fibrillation;
5. Judged to have poor response to loop diuretics before randomisation: presence of symptoms and signs of fluid retention after the administration of a cumulative dose of oral or intravenous loop diuretics equivalent to oral furosemide ≥40 mg (or equivalent doses of other loop diuretics#) within the past 12 hours.

Exclusion Criteria:

1. Myocardial infarction, stroke or transient cerebral ischaemic attack, sustained ventricular tachycardia or ventricular fibrillation within 1 month prior to screening; or severe infection, major trauma or undergoing major or medium-sized surgery within 1 month prior to screening;
2. Coronary revascularisation (percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG)), atrial flutter/fibrillation ablation, pacemaker implantation, valve repair/replacement, carotid or peripheral artery revascularisation, cardiac mechanical assist device therapy, heart transplantation within 1 month prior to screening or planned during the trial; or current severe coronary artery disease or cerebrovascular disease without revascularisation;
3. Fluid retention symptoms and signs judged by the investigator to be caused by non-cardiac diseases; or concomitant conditions causing dyspnoea or fluid retention, such as acute exacerbation of chronic obstructive pulmonary disease, pulmonary heart disease, severe anaemia, decompensated liver cirrhosis, nephrotic syndrome, etc.;
4. Acute heart failure requiring primary correction of the underlying cause as determined by the investigator, due to the following conditions: coronary atherosclerotic heart disease requiring revascularisation, active myocarditis, constrictive pericarditis, cardiac tamponade, complex congenital heart disease, untreated severe primary valvular heart disease, etc.;
5. Previously diagnosed hypertrophic cardiomyopathy (obstructive or non-obstructive), amyloid cardiomyopathy;
6. Use of cardiac mechanical assist device at the time of screening;
7. Hypovolaemia or peripheral perfusion insufficiency at the time of screening, requiring vasoactive drugs, positive inotropic drugs or volume expansion therapy as assessed by the investigator;
8. Anuria at the time of screening; or urinary difficulties caused by urinary tract obstruction, stones or tumours;
9. Unable to perceive thirst at the time of screening, or any reason causing difficulty in fluid intake;
10. Unable to complete weight measurement or urine collection;
11. Consciousness impairment at the time of screening, or hepatic encephalopathy at the time of screening or a history of hepatic encephalopathy;
12. Poorly controlled diabetes at the time of screening, with fasting blood glucose ≥11.1mmol/L;
13. Any organ system malignancy within the last 5 years requiring ongoing treatment such as chemotherapy, radiotherapy, endocrine therapy, targeted therapy, etc.;
14. History of drug abuse or substance use within 1 year prior to screening.
15. Body mass index (BMI) less than 18.5 or greater than 35 kg/m2;
16. Symptomatic hypotension and/or systolic blood pressure <90 mmHg;
17. Estimated glomerular filtration rate (eGFR) <15 mL/min/1.73 m2 (calculated using the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI2009] formula based on serum creatinine), or undergoing/planned for haemodialysis or ultrafiltration therapy;
18. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥3× the upper limit of normal (ULN), except if assessed by the investigator as due to heart failure;
19. Serum sodium > ULN or <130 mmol/L;
20. Serum potassium > ULN or serum potassium still < lower limit of normal (LLN) after treatment;
21. Concurrent active hepatitis B (hepatitis B surface antigen [HBsAg] positive and peripheral blood hepatitis B virus DNA positive) or any one of human immunodeficiency virus antibodies (HIV-Ab), Treponema pallidum antibodies (Anti-TP), hepatitis C virus antibodies (HCV-Ab) positive.
22. Known or suspected allergy to tolvaptan tablets, OPC-61815 injection, or HRS-9057 injection components;
23. Participation in any drug or medical device clinical trial within 3 months prior to screening, defined as: signing the informed consent and using the investigational product (excluding placebo) or investigational medical device; or still within 5 half-lives of the investigational drug (whichever is longer);
24. Use of tolvaptan tablets, OPC-61815 injection, or thiazide diuretics (including combination formulations) within 5 half-lives before dosing;
25. Use of drugs that may affect tolvaptan metabolism within 2 weeks or 5 half-lives before dosing (whichever is longer), includin

    ⅰ strong or moderate CYP3A inhibitors: ketoconazole or other strong CYP3A inhibitors (such as clarithromycin, itraconazole, telithromycin, saquinavir, nelfinavir, ritonavir, nefazodone), moderate CYP3A inhibitors (such as erythromycin, fluconazole, aprepitant, diltiazem, verapamil, delavirdine);

    ⅱ CYP3A inducers: rifampicin or other inducers (such as rifabutin, rifapentine, barbiturates, phenytoin, carbamazepine, forsythia);

    ⅲ P-glycoprotein inhibitors: such as cyclosporine;
26. History of blood donation or blood loss ≥400 mL within 3 months prior to screening, or blood transfusion within 2 months;
27. Participants with mental incapacity or speech disorders, or unable to fully understand or participate in the trial process, or unable to fully understand potential adverse reactions during the study;
28. Pregnant or breastfeeding women, or participants of childbearing potential unwilling to use protocol-specified contraception during the trial and for 1 week after the last dose;
29. As judged by the investigator, any condition affecting participant safety or otherwise interfering with the evaluation of trial results (medical, psychological, social, or geographical factors, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2025-12-31 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Absolute change in weight from baseline on day 8 | within 8 days after the start of administration

SECONDARY OUTCOMES:
Absolute change in body weight from baseline at each visit during treatment | At each visit during treatment，within 8 days after the start of administration
The proportion of participants requiring remedial treatment during therapy as defined by the protocol | after the last case has left the group，within 1years after the first case in
Total dose of loop diuretics during treatment | within 8 days after the start of administration
The incidence and severity of any adverse events (AEs), adverse events of special interest (AESIs), and serious adverse events (SAEs) occurring after any treatment | within 8 days after the start of administration
Incidence of hypernatraemia during treatment | within 8 days after the start of administration
Proportion of participants who experienced hypovolaemic events during treatment and needed to discontinue the trial medication | within 8 days after the start of administration
Detection indicators: concentrations of HRS-9057, tolvaptan and other major metabolites (if applicable) | within 8 days after the start of administration

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided